CLINICAL TRIAL: NCT00678925
Title: Supplemental Choline and Neurodevelopment in Humans
Brief Title: Supplemental Choline and Brain Development in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Gerber Foundation (Other)
Collaborators: Egg Nutrition Center (Other)
Responsible Party: Steve H. Zeisel, MD, PhD, University of North Carolina at Chapel Hill
Organization: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 04-1752 (completed)
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
MeSH Terms: interventions — Phosphatidylcholines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Choline supplement given from 18-weeks pregnancy through 90 days postpartum
  Interventions: Dietary Supplement: Phosphatidylcholine
- 2 (Placebo Comparator): Placebo capsules given from 18 weeks pregnancy through 90 days postpartum
  Interventions: Dietary Supplement: Corn oil placebo

INTERVENTIONS:
Dietary Supplement: Phosphatidylcholine — 850 mg per day from 18 weeks pregnancy through 90 days postpartum
  Other Names: PhosChol
  Arms: 1
Dietary Supplement: Corn oil placebo — Placebo capsules containing corn oil given from 18 weeks pregnancy through 90 days postpartum
  Arms: 2

SUMMARY:
Studies have shown that choline is a necessary part of the human diet. Choline is important in making membranes for all the cells in the body, and for making chemicals that are responsible for nerve function. Studies have also shown that choline improves memory of rats when they are given choline at early stages in their lives. The purpose of this study is to find out whether choline supplementation (provided as a choline dietary supplement) in pregnant women will improve memory function of their babies after they are born.

In this study, we hypothesize that high dietary choline consumption during pregnancy and lactation will:

1. Increase maternal choline concentration in plasma
2. Increase breast milk choline concentration
3. Enhance memory performance in the children born of supplemented mothers

DETAILED DESCRIPTION:
The development of brain during critical periods in embryogenesis is vulnerable to changes in diet, specifically changes in choline intake. Babies born of mothers eating more choline are smarter on memory testing. These effects of dietary choline have been repeatedly demonstrated in rodent models in a series of studies funded by the NIH during the last eight years. Specifically, prenatal choline supplementation in rats facilitates cognitive function and visuospatial memory, whereas choline deficiency impairs divided attention and accelerates the age-related decline in temporal processing. There are two sensitive periods in rat brain development during which treatment with choline produces long-lasting enhancement of spatial memory that is lifelong. The first occurs during embryonic days 12-17 (rats give birth on day 21) and the second, during postnatal days 16-30. Choline supplementation during these critical periods elicits a major improvement in memory performance at all stages of training on a 12-arm radial maze. These changes in memory are correlated with decreases in the threshold for induction of long-term potentiation and with biochemical changes. Choline supplementation in pregnant rats decreases choline acetyltransferase activity and increases phospholipase D (PLD) activity in the hippocampus of offspring. Also, it increases the size of the cell body of cholinergic neurons. In contrast choline deficiency increases the activity of cholinergic system, but does not affect the basal level of PLD activity in hippocampus. These long-lasting functional, anatomical, and biochemical alterations may be related to the changes in neurogenesis and differentiation in fetal hippocampus and septum, areas of brain that are important for normal spatial learning and memory.

It is not known if these findings in rodents are likely to be true in humans, as human and rat brains mature at different rates. Moreover, rat brain is comparatively more mature at birth than is the human brain, but in humans hippocampal development may start around 20 weeks gestation and continue for months after birth. However, everything we know about brain development tells us that the processes seen in rodents are the same as those that occur in the developing human brain. For this reason, it is extremely likely that the robust effects we observe for choline in rodent brain have importance in the human. The research is the first major study in humans to determine whether maternal diet and diet during the baby's first year influences brain function.

ELIGIBILITY:
Inclusion Criteria:

* Less than 18 weeks pregnant
* Intends to breastfeed
* Receives regular prenatal care
* Takes a prenatal vitamin

Exclusion Criteria:

* Uses tobacco or illicit drugs
* Consumes alcohol
* History of chronic illness
* History of allergy to soy or corn
* Difficulty swallowing large capsules
* BMI <18 or >35
* Pregnant with more than 1 fetus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2004-12; Primary Completion 2007-12 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Infant working memory | 10 months & 12 months of age

SECONDARY OUTCOMES:
Breast milk choline concentration | 45 & 90 days postpartum
Plasma choline concentrations | 20 & 30 wks pregnancy, 45 & 90 days postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Cheatham CL, Goldman BD, Fischer LM, da Costa KA, Reznick JS, Zeisel SH. Phosphatidylcholine supplementation in pregnant women consuming moderate-choline diets does not enhance infant cognitive function: a randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2012 Dec;96(6):1465-72. doi: 10.3945/ajcn.112.037184. Epub 2012 Nov 7. PMID 23134891
- [Derived] Fischer LM, da Costa KA, Galanko J, Sha W, Stephenson B, Vick J, Zeisel SH. Choline intake and genetic polymorphisms influence choline metabolite concentrations in human breast milk and plasma. Am J Clin Nutr. 2010 Aug;92(2):336-46. doi: 10.3945/ajcn.2010.29459. Epub 2010 Jun 9. PMID 20534746